CLINICAL TRIAL: NCT03429751
Title: Ultrasound Lung Evaluation of Different Fluid Management Protocols in Patients Undergoing Laparoscopic Hysterectomy.
Brief Title: Ultrasound Lung Fluid Responsiveness During Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mazy (Other)
Responsible Party: Sponsor-Investigator, Alaa Mazy, associate professor of anesthesia and surgical intensive care, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MS/16.06.76
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Fluid Overload
Keywords: lung ultrasound, fluid, hysterectomy, B lines
MeSH Terms: conditions — Edema | interventions — Crystalloid Solutions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal fluid group (Experimental): received 30 ml/Kg/h crystalloid for maximum 3 hours.
  Interventions: Drug: 30 ml/Kg/h crystalloid
- Restrictive fluid group (Active Comparator): received 10 ml /Kg/h crystalloids for maximum 3 hours.
  Interventions: Drug: 10 ml/Kg/h crystalloid

INTERVENTIONS:
Drug: 30 ml/Kg/h crystalloid — Lung ultrasound 8 region assessment using curvilinear 2 to 5 megahertz prob after receiving 30 ml/Kg/h crystalloid in addition to losses for maximum 3 hours.
  Arms: Liberal fluid group
Drug: 10 ml/Kg/h crystalloid — Lung ultrasound 8 region assessment using curvilinear 2 to 5 megahertz prob after receiving 10 ml/Kg/h crystalloid in addition to losses for maximum 3 hours.
  Arms: Restrictive fluid group

SUMMARY:
Bedside lung ultrasound can detect pulmonary congestion by detecting the appearance of B-lines. Pulmonary edema may occur even without cardiomyopathy or heart failure, especially after excessive fluid administration. B-lines have been acknowledged as sonographic signs of pulmonary interstitial and alveolar edema in critical and emergency care. Limited scientific evidence on optimal intraoperative fluid management has resulted in large variations of administered fluid regimens in daily practice. The restricted perioperative intravenous fluid regimen reduces complications after elective surgeries, however other studies had shown that intraoperative liberal fluid administration improves postoperative organ functions and recovery and shortens hospital stay after elective surgeries.

DETAILED DESCRIPTION:
A review of patients undergoing major abdominal surgery, excluding high-risk patients, compared liberal and restrictive ﬂuid regimens; concluded that it is difficult to define 'liberal' or 'restrictive' protocols in clinical practice. patients undergoing moderate-risk surgery seem to benefit from the more liberal fluid administration, while patients undergoing high-risk or major surgery seem to benefit from restrictive or conservative strategies. Lung ultrasound used for comparison between liberal and restrictive fluid therapy in laparoscopic hysterectomy patients by detecting the B-lines intraoperatively or immediately postoperatively. The aim is to evaluate the lung ultrasound as a guide for intraoperative fluid management, being an index for increased extravascular lung water (ECLW). This operation is a moderately complex procedure that implies the Trendelenburg position. This position - in addition to liberal fluids - will increase venous return and increase the challenge on the cardiac muscle under anesthesia in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled for an elective laparoscopic hysterectomy.
* American society of anesthesiologists status I-II.

Exclusion Criteria:

* Patient refusal.
* Severe cardiac insufficiency (New York Heart Association IV, myocardial infarction 3 months).
* Valvular heart diseases.
* Renal insufficiency (GFR<60 ml/kg/1.73m2).
* Hepatic insufficiency (Albumin less than 3).
* Patient with previous or current history of pulmonary disease.
* History of allergy to anesthetic drugs.
* Obese patients (BMI>30).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Endometrial carcinoma patients scheduled for an abdominal hysterectomy.
Enrollment: 48 (Actual)
Dates: Start 2016-07-10 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
The rate of lung ultrasound B lines appearance. | 5 minutes after the end of surgery.
  Three or more comet lines appearance in a lung field. Two or more positive regions per side suggested a B-pattern. B -lines are defined as discrete laser-like vertical hyper-echoic artifacts that arise from the pleura line extend to the bottom of the screen without fading and move synchronously with lung sliding.

SECONDARY OUTCOMES:
The total volume of crystalloid infusion. | Intraoperative.
  milliliter
The total volume of blood transfusion. | Intraoperative.
  milliliter
The amount of blood loss. | Intraoperative.
  milliliter, estimated from the weight of swaps and suction bottles.
The duration of surgery. | intraoperative.
  minutes. from the time of induction of anesthesia till extubation time.
Central venous pressure | Basal 15 minutes preoperative, intraoperative at 15, 30, 45, 60, 90, 120, 150, 180 minutes.
  centimeter water.
Mean blood pressure | Basal 15 minutes preoperative, intraoperative at 15, 30, 45, 60, 90, 120, 150, 180 minutes.
  millimeter mercury.
Heart rate. | Basal 15 minutes preoperative, intraoperative at 15, 30, 45, 60, 90, 120, 150, 180 minutes.
  Beats per minute.
Peripheral oxygen saturation. | Basal 15 minutes preoperative, intraoperative at 15, 30, 45, 60, 90, 120, 150, 180 minutes.
  percent.
Hourly urine output. | intraoperative,
  milliliter,
Arterial blood gases. | 15 minutes preoperative, 15 minutes postoperative.
  for arterial oxygen and carbon dioxide tensions in millimeter mercury, base excess level in millimole per liter.
Serum sodium level. | 15 minutes preoperative, 15 minutes postoperative.
  millimole per liter.
Serum potassium level. | 15 minutes preoperative, 15 minutes postoperative.
  millimole per liter.
Hemoglobin level. | 15 minutes preoperative, 15 minutes postoperative.
  milligram per deciliter.
Hematocrit value. | 15 minutes preoperative, 15 minutes postoperative.
  percent.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Center Mansoura University., Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided